CLINICAL TRIAL: NCT03069248
Title: Treatment of Follicular Non-Hodgkin's Lymphoma With High Dose Therapy and Stem Cell Support Followed by Consolidative Immunotherapy With Rituximab and Alpha Interferon
Brief Title: Treatment of Follicular Lymphoma With High Dose Therapy and Stem Cell Support Followed by Rituximab and Alpha Interferon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Neil Berinstein, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 089-2000
Record Dates: First submitted 2017-02-17; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): Salvage treatment with CHOP or DHAP followed by high dose therapy and stem cell support prior to consolidative immunotherapy with Rituximab and Alpha interferon.
  .
  Interventions: Drug: Rituximab; Drug: Alpha Interferon

INTERVENTIONS:
Drug: Rituximab
Drug: Alpha Interferon

SUMMARY:
This is a non-comparative, prospective, non-randomized single centre phase II clinical trial of Rituximab and alpha interferon immunotherapy following autologous stem cell transplant in patients with relapsed follicular lymphoma conducted at Toronto Sunnybrook Regional Cancer Centre/Sunnybrook and Women's Health Sciences Centre.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1-2 relapses of WHO Classification follicle centre NHL grade 1-2/3. Patients must have achieved at least a PR to previous treatment.
* Central pathology review before registration
* Ann Arbor stage III or IV
* Measurable disease: defined as clinically or radiologically documented disease with at least one site bidimensionally measurable using clinical exam, CT or MRI performed in the 3 weeks prior to study enrollment.
* ECOG performance status of <2.
* Patients may have received not more than 1 prior course (4 infusions) of rituximab. Timing of rituximab must exceed 12 months prior to registration. Patients must have demonstrated at least a PR to rituximab if previously administered.
* Patient consent according to institutional and university human experimentation committee requirements
* Adequate Renal, hepatic and hematopoietic function test unless the abnormal values are thought to be due to involvement with lymphoma as defined by:

Hb> 85 ANC >1000/mm3 Platelets >100,000/mm3 Serum/Total Bilirubin >=2 SI units AST/ALT <2x Upper Limit of Normal

Exclusion Criteria:

* Positive serology for HIV
* Uncontrolled Infection
* Pregnancy
* CNS Metastases
* History of Psychiatric Disorder
* Other Malignancy (except nonmelanoma skin cancer)
* Serious non-malignant disease (e.g., congestive heart failure, or active uncontrolled bacterial, viral, or fungal infections), or other conditions, which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives.
* Major surgery, other than diagnostic surgery, within four weeks.
* Presence of anti-murine antibody (HAMA) reactivity. These laboratory results must be available prior to receiving treatment for those patients
* who have received prior murine proteins or patients who have allergies to murine proteins.
* New York Heart Association Class III or IV heart disease (see Appendix H, Clinical Evaluation of Functional Capacity of Patients with Heart Disease in Relation to Ordinary Physical Activity) or myocardial infarction within the past six months.
* Treatment with an investigational drug within 30 days or five half-lives (of the study drug with the longest half-life) prior to entry into the study, which ever is longer.
* Previous chemotherapy, immunotherapy, radiotherapy, or investigational therapy for the treatment of other malignancy except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix within the last 5 years.
* History of allergic reactions to compounds chemically related to Rituximab.
* Refusal to practice contraception if of reproductive potential.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-06-01 (Actual); Primary Completion 2009-09-17 (Actual); Study Completion 2009-09-17 (Actual)

PRIMARY OUTCOMES:
Survival (Overall survival) | From date of randomization until date of death or last follow-up, whichever comes first, assessed up to 116 months
  Overall survival
Survival (Progression free survival) | From date of randomization until date of relapse or disease progression, assessed up to 116 months
  Progression free survival

SECONDARY OUTCOMES:
Toxicities (Possible transplant-related adverse events) | assessed semi-annually, from date of enrollment up to 116 months
  Possible transplant-related adverse events such as secondary malignancies, hypogammaglobulinemia, and pulmonary fibrosis
Minimal Residual Disease | assessed semi-annually, from date of enrollment up to 116 months
  Occult disease by PCR analysis of the t(14;18) or of patient specific V(D)J rearrangements in peripheral blood, bone marrow and stem cell graft collections.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Berinstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No